CLINICAL TRIAL: NCT00643253
Title: Provider Approaches to Improved Rates of Infant Nutrition and Growth Study
Acronym: PAIRINGS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Albert Einstein College of Medicine (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Karen Bonuck, Professor, Albert Einstein College of Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 2007-490-000; 1P60MD00516
Record Dates: First submitted 2008-03-24; First posted 2008-03-26 (Estimated); Last update posted 2013-07-11 (Estimated); Status verified 2013-07

CONDITIONS: Breastfeeding
Keywords: exclusive breastfeeding; breastfeeding promotion; health promotion
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Receipt of behavioral interventions to encourage breastfeeding.
  Interventions: Behavioral: LC and Electronic Prompt
- 2 (No Intervention): Standard of Care

INTERVENTIONS:
Behavioral: LC and Electronic Prompt — Women will receive: a) International Board of Certified Lactation Consultant (IBCLC) education/counseling during the pre-natal, intra-partum and post-hospital discharge period to promote early and continued exclusive breastfeeding. The protocol specifies 2 prenatal meetings, a hospital visit, and a home visit if indicated and accepted, and; b) Electronic Medical Record Prompts- will appear on the prenatal record 5 times throughout the pregnancy. They are brief discussion points re breastfeeding that the provider is asked to raise with their patients.
  Other Names: breastfeeding promotion; lactation consultant intervention; electronic health promotion
  Arms: 1

SUMMARY:
We will conduct a randomized, controlled trial of routine, pre-natal care practice-site based pre- and post-natal breastfeeding promotion interventions in low-income minority women, with stratification for maternal country of origin. Our primary outcome measure is breastfeeding duration and extent, i.e. "intensity." Our secondary outcomes measures are: a) infant weight, and b) participant/ provider experiences of the intervention.

The Provider Approaches to Improved Rates of Infant Nutrition & Growth Study (PAIRINGS) trial randomizes women to a Prenatal Care Provider (PNC) + Lactation Consultant (LC) intervention, or Control group. The PNCs will use a brief, computer prompted protocol throughout pregnancy and at follow-up of maternal-infant dyads. The LC will meet women, one-on-one while pregnant, at daily hospital rounds, during well-infant care and (as needed) home visits. Post-partum interviews at 1,3 and 6 months will collect infant feeding data.

Primary Outcomes (Hypotheses): Breastfeeding

1. Breastfeeding Intensity at 1,3, and 6 Months- There will be significant differences, by treatment group, in BF intensity. Intensity will be assessed via 7 day recall of the frequency of breastmilk feedings vs. other liquids and solids.
2. Exclusive Breastfeeding at 1,3, and 6 Months- There will be significant differences, by treatment group, in the rate of exclusive BF.

   Secondary Outcomes (Hypotheses): Infant Growth
3. Weight-for-Length, by Breastfeeding Intensity: There will be a significant association between BF intensity and weight-for-length z scores at 4,6,9, and 12 month well-child visits.
4. Weight Gain, by Breastfeeding Intensity: There will be a significant association between BF intensity and weight gain from the 4th -12th month of age.
5. Weight-for-Length, by Treatment Group: There will be a significant association between treatment group and weight-for-length z scores at 4,6,9, and 12 month well-child visits
6. Weight Gain, by Treatment Group: There will be a significant association between treatment group and weight gain from the 4th - 12th month of age.

ELIGIBILITY:
Inclusion Criteria:

* 12-30 weeks pregnant
* receives prenatal care at Centennial women's center of Montefiore Medical Center
* English or Spanish speaking

Exclusion Criteria:

* pregnant with multiples
* breastfeeding contra-indicated

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 299 (Actual)
Dates: Start 2008-03; Primary Completion 2012-09 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Breastfeeding intensity at 1,3, and 6 months | 1,3, and 6 months after birth of the baby

SECONDARY OUTCOMES:
Infant growth by treatment group and breastfeeding intensity | Assessed when baby is 1,3, and 6 months of age

CONTACTS AND LOCATIONS:
Overall Officials: Karen A. Bonuck, PhD, Principal Investigator — Albert Einstein College of Medicine
Locations (1):
- Dept of Obstetrics, Gynecology, and Women's Health/Centennial Building/Montefiore Medical Center, The Bronx, New York, United States

REFERENCES:
- [Derived] Bonuck K, Stuebe A, Barnett J, Labbok MH, Fletcher J, Bernstein PS. Effect of primary care intervention on breastfeeding duration and intensity. Am J Public Health. 2014 Feb;104 Suppl 1(Suppl 1):S119-27. doi: 10.2105/AJPH.2013.301360. Epub 2013 Dec 19. PMID 24354834
- [Derived] Andaya E, Bonuck K, Barnett J, Lischewski-Goel J. Perceptions of primary care-based breastfeeding promotion interventions: qualitative analysis of randomized controlled trial participant interviews. Breastfeed Med. 2012 Dec;7(6):417-22. doi: 10.1089/bfm.2011.0151. Epub 2012 May 23. PMID 22621223